CLINICAL TRIAL: NCT03344224
Title: The Relationship of Pre-operative Blood Lipid Level and Post-operative Major Adverse Cardiac Event Occurence
Brief Title: Pre-operative Blood Lipid Level and Post-operative Major Adverse Cardiac Event
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator,, Peking University First Hospital
Other Study IDs: LMACE
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Lipid Metabolism Disorders; Postoperative Complications
MeSH Terms: conditions — Lipid Metabolism Disorders; Postoperative Complications | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal blood lipid/protein group
  Interventions: Diagnostic Test: laboratory test
- abnormal blood lipid/protein group
  Interventions: Diagnostic Test: laboratory test

INTERVENTIONS:
Diagnostic Test: laboratory test — laboratory test

SUMMARY:
Whether the pre-operative blood lipid level and post-operative cardiovascular events is associated is unknown. This study is to find out the main blood lipid and relative protein level change and the post-operative cardiovascular events occurrence.

DETAILED DESCRIPTION:
The participants collected data from their hospital.Patients under going non-cardiac surgery were collected. Data of Triglycerides, cholesterol, Low-density lipoprotein and High-density lipoprotein were collected perioperatively. The postoperative major cardiovascular and cerebral events were also identified and collected. Other data including perioperative information and surgeries and anesthesia data were gathered.

Logistic regression models were built and selected. Independent risk factors relative to postoperative major cardiovascular and cerebral events were screened and identified. different levels of Triglycerides, cholesterol, Low-density lipoprotein and High-density lipoprotein were analysed.

ELIGIBILITY:
Inclusion Criteria:

* non-cardiac surgery patients with preoperative blood lipid tests

Exclusion Criteria:

* electronic records missing or peri-operative data missing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult non-cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
cardiovascular events | 30 days postoperatively
  such as acute myocardial infarction

REFERENCES:
- [Background] Leardi S, Altilia F, Delmonaco S, Cianca G, Pietroletti R, Simi M. [Blood levels of cholesterol and postoperative septic complications]. Ann Ital Chir. 2000 Mar-Apr;71(2):233-7. Italian. PMID 10920496